CLINICAL TRIAL: NCT03622034
Title: Knee Posterior Femoral Condylar Offset and Tibial Slope of the Egyptian Population
Acronym: knee
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MBMady, resident of orthopedics and trauma surgery, Assiut University
Other Study IDs: knee measures
Record Dates: First submitted 2018-07-28; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Changes in Knee Measurements Between Egyptian and Western Population
Keywords: knee features; ethnic changes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: posterior condylar offset measurement — the tangent to the medial tibial plateau is considered to be the proximal reference line. This is the line connecting the highest anterior and posterior points of the medial plateau. The second reference is the axis of the tibia, defined as a line through the middle of the shaft at 10 and 20 cm. The angle between these two lines is the tibial slope
  Other Names: tibial slope measurement

SUMMARY:
this study is to compare the posterior condylar offset , posterior condylar offset ratio and tibial slope of Egyptian population with Asian and Western results.These results may be important to examine if contemporary total knee arthroplasty components match the anatomy of Egyptian populations or they are significantly different with the need of different prosthesis designs and geometrics.

DETAILED DESCRIPTION:
Lateral knee x rays will be collected from the registry system of Assiut University Hospital through Paxera pacs system . Posterior condylar offset, posterior condylar offset ratio and tibial slope will be measured from the x rays.

In the sagittal plane, the femoral long axis will be drawn with equal distance to the anterior-posterior edges of the femoral shaft. One line will be drawn parallel to the anterior femoral shaft cortex and another parallel to the posterior femoral shaft cortex. A third line will be drawn parallel to the posterior femoral shaft cortex line, but tangent to the most posterior femoral condyles to represent the posterior condylar tangent line. The anterior-posterior dimension of the distal femur is defined as the distance between the anterior femoral shaft cortex line and the posterior femoral condyle tangent line . The posterior femoral condyle offset (PCO) is determined as the distance between the posterior femoral shaft cortex line and the posterior femoral condyle line, that is noted as PCO .The posterior femoral condyle offset ratio (PCOR) is calculated as the ratio of the posterior femoral condyle offset and the anterior-posterior dimension of the distal femur, i.e., PCO/ACP.

Tibial slope will be measured as follows; the tangent to the medial tibial plateau is considered to be the proximal reference line. This is the line connecting the highest anterior and posterior points of the medial plateau. The second reference is the axis of the tibia, defined as a line through the middle of the shaft at 10 and 20 cm. The angle between these two lines is the tibial slope.

Data of the cases will be collected as name, age and gender. The results will be collected and will be compared with those of Asian and Western results. These results may be important to examine if contemporary TKA components match the anatomy of Egyptian populations or they are significantly different with the need of different prosthesis designs and geometrics.

ELIGIBILITY:
Inclusion Criteria:

* Proper lateral knee x ray of adult cases

Exclusion Criteria:

* 1. Improper x ray projection
* 2. Retained hardware
* 3. Malunited distal or upper tibia fracture

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all adult cases who have proper lateral knee x ray on the registery system of Assiut University Hospital , will be collected. These x rays will be used in this study as posterior condylar offset, posterior condylar offset ratio and tibial slope will be measured on these x rays
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure posterior condylar offset in the Egyptian population | one year
  posterior condylar offset will be measured in a sample of the egyptian people to get the mean measure of posterior condylar offset in the egyptian people

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwak DS, Tao QB, Todo M, Jeon I. Determination of representative dimension parameter values of Korean knee joints for knee joint implant design. Proc Inst Mech Eng H. 2012 May;226(5):368-76. doi: 10.1177/0954411912442025. PMID 22720389
- [Background] Mahfouz M, Abdel Fatah EE, Bowers LS, Scuderi G. Three-dimensional morphology of the knee reveals ethnic differences. Clin Orthop Relat Res. 2012 Jan;470(1):172-85. doi: 10.1007/s11999-011-2089-2. PMID 21948324
- [Background] Bellemans J, Carpentier K, Vandenneucker H, Vanlauwe J, Victor J. The John Insall Award: Both morphotype and gender influence the shape of the knee in patients undergoing TKA. Clin Orthop Relat Res. 2010 Jan;468(1):29-36. doi: 10.1007/s11999-009-1016-2. Epub 2009 Aug 8. PMID 19669385
- [Background] Conley S, Rosenberg A, Crowninshield R. The female knee: anatomic variations. J Am Acad Orthop Surg. 2007;15 Suppl 1:S31-6. doi: 10.5435/00124635-200700001-00009. PMID 17766787
- [Background] DiBennardo R, Taylor JV. Sex assessment of the femur: a test of a new method. Am J Phys Anthropol. 1979 May;50(4):635-7. doi: 10.1002/ajpa.1330500415. PMID 464035
- [Background] Leszko F, Hovinga KR, Lerner AL, Komistek RD, Mahfouz MR. In vivo normal knee kinematics: is ethnicity or gender an influencing factor? Clin Orthop Relat Res. 2011 Jan;469(1):95-106. doi: 10.1007/s11999-010-1517-z. PMID 20814773
- [Derived] Abdelnasser MK, Abdelhameed MA, Bassem M, Adam MF, Bakr HM, Khalifa YE. Sexual dimorphism of the posterior condylar offset of the femur and the medial posterior slope of the tibia in non-arthritic knees of Egyptian adults: an MRI study. J Orthop Surg Res. 2023 May 12;18(1):353. doi: 10.1186/s13018-023-03833-2. PMID 37173701
- [Derived] Abdelnasser MK, Khalifa AA, Bassem M, Abdelhameed MA, Adam MF, Bakr HM, Khalifa YE. Anthropometric measurements of non-arthritic knees in an Egyptian population: an MRI-based study. J Orthop Surg Res. 2021 Sep 8;16(1):552. doi: 10.1186/s13018-021-02708-8. PMID 34496904